CLINICAL TRIAL: NCT03195556
Title: Augmentation of Limb Perfusion With Contrast Ultrasound
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Jonathan R. Lindner, MD, Professor, Oregon Health and Science University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00017343
Record Dates: First submitted 2017-06-16; First posted 2017-06-22 (Actual); Last update posted 2018-08-23 (Actual); Status verified 2018-08

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Healthy subjects (Experimental): Low-power contrast ultrasound perfusion imaging and measurement of ABI and TBI will be performed before and after a 15 min high-power ultrasound cavitation therapy with intermittent ultrasound and intravenous infusion of microbubbles.
  Interventions: Device: Ultrasound
- Peripheral Artery Disease (Experimental): Low-power contrast ultrasound perfusion imaging and measurement of ABI and TBI will be performed before and after a 15 min high-power ultrasound cavitation therapy with intermittent ultrasound and intravenous infusion of microbubbles.
  Interventions: Device: Ultrasound

INTERVENTIONS:
Device: Ultrasound — Ultrasound exposure of Definity microbubbles infused over 10 min. Ultrasound administered at 1.3 MHz, mechanical index of 1.3, and pulsing interval of 10 s.
  Other Names: Contrast ultrasound

SUMMARY:
Our laboratory has discovered that ultrasound (US) imaging together with clinically approved microbubble ultrasound contrast agents can augment limb tissue perfusion. These observations have been made in mice with and without peripheral artery disease (PAD), and also in humans where high power contrast enhanced ultrasound (CEU) was used to measure perfusion but was found also to augment perfusion by almost 2-fold. The latter human studies were performed with ultrasound protocols designed for perfusion imaging and not for flow augmentation. In this study, we will measure the degree to which limb perfusion is augmented with specific therapeutic CEU settings that are still within the FDA-approved limits with regards to US power and contrast dosing.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 y.o.
* For PAD subjects: known history of unilateral or bilateral PAD diagnosed by reduced ankle-brachial index or angiography and a Rutherford symptom class of 4-6.

Exclusion Criteria:

1. Major medical illness other than PAD affecting the limb (muscle disease, blood diseases that influence flow or rheology, severe heart failure [NYHA class IV or LVEF <30%]).
2. Pregnant or lactating females
3. Hypersensitivity to any ultrasound contrast agent
4. Known atrial septal defect or large right to left shunt.
5. Hemodynamic instability (hypotension with systolic BP <90 mm Hg, need for vasopressors)
6. Evidence for ongoing myocardial ischemia
7. For normal controls, any known structural non-arrhythmic cardiovascular disease (coronary artery disease, heart failure, moderate or greater valve disease).

Ages: 19 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-06-18 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Change in blood flow at 10 min | 10 min post-therapeutic ultrasound cavitation.
  Change in blood flow in calf skeletal muscle
Change in blood flow at 60 min | 60 min post-therapeutic ultrasound cavitation
  Change in blood flow in calf skeletal muscle

CONTACTS AND LOCATIONS:
Locations (1):
- OHSU, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mason OR, Davidson BP, Sheeran P, Muller M, Hodovan JM, Sutton J, Powers J, Lindner JR. Augmentation of Tissue Perfusion in Patients With Peripheral Artery Disease Using Microbubble Cavitation. JACC Cardiovasc Imaging. 2020 Mar;13(3):641-651. doi: 10.1016/j.jcmg.2019.06.012. Epub 2019 Aug 14. PMID 31422129